CLINICAL TRIAL: NCT03021876
Title: L-carnitine Corrects Ammonia Metabolism in Hepatectomized Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Division Manager, Kochi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAMP study
Record Dates: First submitted 2016-03-12; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Ammonia Metabolism
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ordinary group (Placebo Comparator): usual intake prior to liver surgery
  Interventions: Other: usual intake
- carnitine group (Active Comparator): treatment with oral L-carnitine, 1500 mg/body per day for 2 weeks prior to liver surgery
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: L-carnitine — treatment with oral L-carnitine, 1500 mg/body per day
  Other Names: Carnitine group
  Arms: carnitine group
Other: usual intake — baseliner
  Other Names: Usual group
  Arms: ordinary group

SUMMARY:
L-carnitine is synthesized from lysine and methionine. Postmortem concentrations of carnitine in liver, muscle, heart, kidney, and brain averaged only one-fourth to one-third those in corresponding tissues of eight normally nourished non-hepatic patients who died after an acute illness of a 1-3-day duration. In the recent years, it has been reported that sirtuin 3 (SIRT3) is protective against acute kidney injury (AKI) and suggest that enhancing SIRT3 to improve mitochondrial dynamics has potential as a strategy for improving outcomes of renal injury. In the current study, it is the first clinical interventional research whether L-carnitine corrects ammonia metabolism associated with liver injury in hepatectomized patients.

ELIGIBILITY:
Inclusion Criteria:

* patients were those surgically treated for hepato-biliary diseases

Exclusion Criteria:

* Patient exclusion criteria included a body weight loss greater than 10% during the six months prior to surgery, the presence of distant metastases, or seriously impaired function of vital organs due to respiratory, renal or heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
postoperative ammonia levels | 3 points; preoperative baseline, postoperative day 1, and day3
  change from preoperative baseline at postoperative day 1 and day3

SECONDARY OUTCOMES:
length of hospitalization after liver resection | up to 24 weeks
  postoperative days

CONTACTS AND LOCATIONS:
Locations (1):
- Kochi Health Sciences Center, Kochi, Kochi, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okabayashi T, Sui K, Mastumoto T, Iwata J, Morita S, Iiyama T, Shimada Y. l-Carnitine Improves Postoperative Liver Function in Hepatectomized Patients. JPEN J Parenter Enteral Nutr. 2020 Jul;44(5):823-830. doi: 10.1002/jpen.1720. Epub 2019 Oct 9. PMID 31599019